CLINICAL TRIAL: NCT04525534
Title: Plasma Concentration of Biological Markers in Placenta Spectrum
Brief Title: Plasma Concentration of Biological Markers in Placenta Accreta Spectrum
Status: Terminated | Type: Observational
Why Stopped: difficulties with enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 261299
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-11

CONDITIONS: Placenta Accreta; Placenta Diseases
MeSH Terms: conditions — Placenta Accreta; Placenta Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood for serum biomarkers and placental micro-particles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Placenta accreta spectrum: Mother-infant dyads with suspected or confirmed diagnosis of placenta accreta spectrum
  Interventions: Other: There is no other intervention, only clinical treatment.
- Phenotypically-matched controlled group: Mother-infant dyads admitted for delivery without placenta accreta spectrum
  Interventions: Other: There is no other intervention, only clinical treatment.

INTERVENTIONS:
Other: There is no other intervention, only clinical treatment. — There is no other intervention, only clinical treatment

SUMMARY:
The purpose of this exploratory study is to determine how well maternal serum biomarkers and placental micro-particles (MP) correlate with placenta accreta spectrum (PAS) at the time of cesarean delivery in women with suspected PAS compared to women without PAS. Our aim is to determine if women with PAS have a unique MP and protein signature at the time of delivery compared with women without PAS.

DETAILED DESCRIPTION:
Maternal blood samples will be taken at various points during the intrapartum period. A healthy group of women admitted for delivery will act as a matched control and will have their blood sampled at similar time points. The primary outcome variables will include the total number of micro-particles, the number of micro-particles from each cell line (platelet, placental, endothelial etc.), and protein markers The knowledge gained from this study has the potential to develop a diagnostic test for PAS with the ability to improve management and outcomes for mother and baby through earlier diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - to 45-years old, inclusive
* Suspected or confirmed PAS or phenotypically matched controls
* Delivery by cesarean section
* Gestational age greater than 28 weeks
* Singleton pregnancy

Exclusion Criteria:

* Intrauterine fetal demise,
* Severe fetal anomalies (infant not expected to survive)
* Emergent cesarean delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mother-infant dyads with suspected or confirmed diagnosis of PAS and healthy mother-infant dyads admitted for cesarean delivery
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Determine the level of placental-derived MPs (Microparticles/mL) | Up to 6 hours
  Determine quantitatively the level of placental-derived MPs which may be altered in 10 subjects with PAS and 10 phenotypically-matched controls.
Identify biomarkers (picogram/mL) | Up to 6 hours
  Determine quantitatively the level of biomarkers which may be altered in 10 subjects with PAS and 10 phenotypically-matched controls.

SECONDARY OUTCOMES:
Is there a correlation between maternal serum total placental MPs and biomarkers to the International Federation of Gynecology and Obstetrics (FIGO) classification for PAS at the time of cesarean delivery. | Up to 6 hours
  Examine the correlation between maternal serum total placental MPs and biomarkers to the FIGO classification

CONTACTS AND LOCATIONS:
Overall Officials: Nadir e Sharawi, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States